CLINICAL TRIAL: NCT01469416
Title: The Effects of Administering Clopidogrel on the Pharmacokinetics of Rosuvastatin in Healthy Volunteers
Brief Title: Drug Interaction Study of Clopidogrel and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11-07522
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: rosuvastatin; clopidogrel; pharmacokinetics; drug interaction; healthy volunteer; drug transporter
MeSH Terms: interventions — Rosuvastatin Calcium; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Rosuvastatin + clopidogrel (Experimental)
  Interventions: Drug: Rosuvastatin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg PO x 1
Drug: Clopidogrel — Clopidogrel 300 mg PO x 1 (30 minutes prior to rosuvastatin dose); Clopidogrel 75 mg PO x 1 (24 hours post-rosuvastatin dose)
  Arms: Rosuvastatin + clopidogrel

SUMMARY:
The purpose of this study is to determine if clopidogrel inhibits hepatic uptake transport of rosuvastatin clinically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, male or female, age 18-65 years old, with no current medical conditions or active diagnoses as determined by the study doctor based on history, physical exam and laboratory evaluations
* Subjects that take no other medications 2 weeks prior to the study and during the time course of the study including prescription medications, over-the-counter medications (except acetaminophen), dietary supplements, or drugs of abuse
* Subjects with a SLCO1B1*1A genotype
* Subjects able to maintain adequate birth control during the study independent of hormonal contraceptive use
* Subjects able to abstain from grapefruit, grapefruit juice, orange juice, caffeinated beverages and/or alcoholic beverages from 3 pm the day before the study to completion of that study day.
* Participants determined to have normal liver and kidney function as measured at baseline
* BMI between 18.5 - 30 kg/m2
* Subjects capable of fasting from food and beverages at least 8 hours prior to medication dosing
* Be able to read, speak, and understand English

Exclusion Criteria:

* Subjects with active medical problems
* Subjects on chronic prescription or OTC medications that cannot be stopped 2 weeks prior to and during the study.
* Subjects incapable of multiple blood draws (HCT <30 mg/dL)
* Subjects with a history of rhabdomyolysis
* Subjects with a history of drug-related myalgias
* Subjects with a history or diagnosis of hemorrhagic tendencies or blood dyscrasias
* Subjects with a history of GI bleed or peptic ulcer disease
* Subjects with a recent history of trauma
* Subjects with a recent history of or upcoming plan of surgery
* Subjects that smoke tobacco or have ongoing alcohol or illegal drug use
* Subjects who are pregnant, lactating, or trying to conceive during the study period
* Subjects allergic to rosuvastatin or clopidogrel or any known component of the medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Area-under-the-concentration curve (AUC) of rosuvastatin | Blood samples collected over a 48 hour period

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of rosuvastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, and 48 hours post-dose
Time to concentration maximum (Tmax) of rosuvastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, and 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, UCSF, San Francisco, California, United States